CLINICAL TRIAL: NCT01980121
Title: Gastric Sonography in the Fasted Term Pregnant Patient for Elective Cesarean Delivery: a Prospective Descriptive Study
Brief Title: Gastric Sonography in the Fasted Term Pregnant Patient for Elective Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 13-08
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Respiratory Aspiration; Pregnancy
Keywords: Respiratory Aspiration; Pregnancy; Ultrasound; Gastric Contents
MeSH Terms: conditions — Respiratory Aspiration | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Term pregnant patients: Term pregnant patients for scheduled elective cesarean section will be examined using a portable ultrasound machine to evaluate gastric contents.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Two-dimensional portable ultrasound unit with a low frequency (2-5 MHz) curved array transducer

SUMMARY:
Food residue in the stomach of patients scheduled to have surgery is considered a major risk factor for pulmonary aspiration of gastric contents. The resulting respiratory compromise after aspiration is associated with significant morbidity and mortality. The risk of pulmonary aspiration is especially important in pregnant women, as they may often require surgery without having observed appropriate fasting. In pregnant patients scheduled for elective surgery, standard preoperative guidelines apply as the general non-pregnant surgical population (8-hour fasting of solid food and 2-hour fasting of clear fluids). A bedside ultrasound assessment of the status of the gastric content and volume would be of great value for the clinician. This technique has recently been shown very promising in fasted non-pregnant patients scheduled for elective surgery. Therefore, it is important to study its feasibility in the pregnant population scheduled for elective Cesarean Delivery.

The investigators hypothesize that no residual solid contents will be found in the gastric sonography, and a small volume of gastric fluid will be observed in the antrum in both supine and right lateral decubitus.

DETAILED DESCRIPTION:
The aim of this prospective study is to provide a qualitative and quantitative description of the sonographic appearance of the gastric antrum in fasted pregnant undergoing elective Cesarean delivery.

The investigators expect that the information obtained from the systematic ultrasonographic qualitative/quantitative assessment of the gastric content may help anesthesiologist to better assess aspiration risk and guide anesthetic and airway management, particularly in pregnant women scheduled for elective Cesarean delivery after standard preoperative fasting guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Non-labouring pregnant women at term (≥ 36 weeks)
* 18 years or older
* ASA Physical Status I-III
* 50-120 kg of weight
* 150 cm of height or taller
* Ability to understand the rationale of the study assessments and to provide signed informed consent
* Written informed consent

Exclusion Criteria:

* Known pre-existing abnormal anatomy of the upper gastrointestinal tract
* History of upper GI tract surgical procedure

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Term pregnant patients who have scheduled elective cesearean sections.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2013-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Qualitative assessment of the antrum of the stomach | 10 minutes
  Patients will be classified as follows; Grade 0: the antrum appears empty on both supine and right lateral decubitus positions; grade 1: gastric fluid is visible on the right lateral decubitus position only, suggesting a small fluid volume; and grade 2: gastric fluid is observed in the antrum in both supine and right lateral decubitus, suggesting a larger fluid volume.

SECONDARY OUTCOMES:
Quantitative assessment of the antrum of the stomach | 10 minutes
  Three consecutive measures of the CSA (cross sectional area) of the antrum will be calculated via the ultrasound machine (free tracing method).

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Arzola, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada